CLINICAL TRIAL: NCT06001060
Title: 1. Study Design 2. Sample Collection 3. Microbial DNA Extraction in Faecal Samples 4. PCR Amplification： 5. Sequencing： 6. HCY Test Principle: 7. Statistical Analysis
Brief Title: Distinct Alterations in Gut Microbiota Composition Among Women of Reproductive Age With Elevated Homocysteine Levels.
Status: Completed | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2023004
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women of reproductive age with elevated homocysteine levels

SUMMARY:
The goal of this observational study is to test the alterations of gut microbiota composition among women of reproductive age with elevated homocysteine levels. The main question it aims to answer is:

• the relationship between gut microbiota composition and recurrent abortion. Participants will provide their stool samples to be detected the composition of gut microbiota. .

Researchers will compare women of reproductive age with normal homocysteine levels to see if any bacteria were involved in recurrent miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* No recent antibiotic treatment

Exclusion Criteria:

* Recently received antibiotics

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: patients or healthy individuals who visited Hangzhou First People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
homocysteine levels | The first day of the trail
  Binding or dimer homocysteine (oxidized form) is reduced to free homocysteine, and then it is catalysed by cysteine β-synthetase (CBS) to react with serine to form cysteine sulfuric acid. Cysteine is then broken down by cysteine β-lyase (CBL) to form homocysteine, pyruvate, and ammonia. Pyruvate is then converted to lactate using lactate dehydrogenase (LDH), where nicotinamide adenine dinucleotide (NADH) is used as a coenzyme. The ratio of NADH to NAD* is directly proportional to the concentration of homocysteine (△ A340 nm).

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes